CLINICAL TRIAL: NCT01194089
Title: A Randomized, Double Blind, Study to Evaluate the Efficacy of Nasal Nicotine Spray to Reduce Post-Operative Opioid Requirements in Nonsmokers in Elective Laparoscopic Bariatric Surgical Patients
Brief Title: Nicotine Administration and Post-operative Opioid Use With Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Toby Weingarten (Other)
Responsible Party: Sponsor-Investigator, Toby Weingarten, Associate Professor of Anesthesiology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-002241
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Pain, Postoperative
Keywords: Nicotine; Postoperative pain; Bariatric surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Nicotine Spray (Active Comparator): 3 mg of nasal nicotine will be administered postoperatively.
  Interventions: Drug: Nasal Nicotine Spray
- Nasal Normal Saline Spray (Placebo Comparator): 1 ml of nasal normal saline spray will be administered postoperatively.
  Interventions: Drug: Nasal Normal Saline Spray

INTERVENTIONS:
Drug: Nasal Nicotine Spray — Single 3 mg dose of nasal nicotine spray
  Other Names: Nicotrol NS
  Arms: Nasal Nicotine Spray
Drug: Nasal Normal Saline Spray — An isotonic solution of sodium chloride 0.65% in deionized water
  Other Names: Rhino-Mist; Salinex; Ocean Nasal Spray
  Arms: Nasal Normal Saline Spray

SUMMARY:
This prospective, randomized, double-blind study will enroll nonsmoking female subjects undergoing laparoscopic bariatric surgery under general anesthesia. The hypothesis of this study is that female nonsmokers who receive nicotine via nasal spray immediately before waking up from anesthesia will need less pain medications 24 hours after the surgery compared to the subjects who receive placebo spray.

DETAILED DESCRIPTION:
Though nicotine is known to be a mild analgesic, its use in the peri-operative period to reduce postoperative opioid requirements has only recently been investigated. In nonsmokers it has been shown to reduce postoperative pain and opioid requirements in both female patients undergoing uterine surgery and male patients undergoing prostatectomy. We have recently confirmed these findings in women undergoing uterine surgery by open, laparoscopic and vaginal approaches. In this study we found a 30% mean reduction of 24 hour postoperative opioid requirements following the administration of a 3 mg dose of nicotine nasal spray. Two previous studies with perioperative transdermal nicotine found that increasing doses of nicotine and increasing serum levels of nicotine were associated with higher rates of nausea. In our study, we found that the administration of nasal nicotine was associated with a transient increase of postoperative nausea and vomiting (PONV), but this was limited to the recovery room (PACU) stay. Two studies of nasal nicotine where antiemetics were prophylactically administered did not report the incidence of nausea. In our study, antiemetics were used as rescue medications only. Thus, it is unclear if the prophylactic administration of anti-emetics would effectively counteract the transient emetogenic effect of a small dose of nasal nicotine.

Laparoscopic bariatric surgery is becoming an increasingly popular treatment of morbid obesity. We recently performed a detailed analysis of postoperative pain and opioid requirements among patients that had this type of surgery and found that among non-smokers severe pain (pain > 7/10 on a 10 point scale) was commonly experienced (35%) despite substantial amount of postoperative opioid use (mean 68 mg oral morphine equivalents) and non-opioid analgesics in the first 24 hours. Because obesity related sleep disorders exceed 70% of patients undergoing bariatric surgery, and those disorders are exacerbated by opioids, potential therapies that could reduce postoperative opioid requirements in these patients have substantial value. Further, delayed nausea often poses a problem for these patients meeting hospital discharge criteria, and opioids used for analgesia aggravates this problem. Thus, the use of nasal nicotine could reduce the amount of opioid these patients require for postoperative analgesia. Combined with aggressive antiemetic prophylaxis against PONV, nasal nicotine could paradoxically and indirectly reduce the incidence of nausea in these patients by decreasing postoperative opioid requirements. The proposed study is a randomized clinical trial examining how nicotine affects recovery of female non-smokers undergoing bariatric surgery from general anesthesia. We will test the hypothesis that nicotine, administered in a nasal spray immediately before emergence from anesthesia, will reduce postoperative opioid requirement and postoperative pain. A secondary outcome is to assess if the routine administration of prophylactic antiemetic therapy prevents increased PONV associated with nicotine administration.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 2-3
* Non-smokers, defined as not smoking (not even a puff) for at least one year preoperatively, and having smoked less than 100 cigarettes throughout their life or remote history of smoking with complete tobacco abstinence (not even a puff) for at least 10 years
* Scheduled for elective laparoscopic bariatric surgery (other than gastric banding or sleeve resection bariatric surgeries as these are outpatient procedures) requiring general anesthesia.

Exclusion Criteria:

* Regular use of opioid medications in the past year, any prior use of sustained release opioid medications, or history of substance abuse with opioids
* History of previous psychiatric hospitalizations
* Allergy to nicotine
* Previous bariatric surgery or previous foregut surgery
* Pregnant or lactating female (per usual surgical routine)
* Contraindications for receiving ketorolac (elevated creatinine)
* Unstable angina, severe uncontrolled hypertension, serious cardiac dysrhythmias (tachyarrhythmias, atrial fibrillation), or vasospastic diseases (Buerger's disease, Raynaud's phenomena)
* Unable to provide informed consent to participate in the study
* Contraindication to the proposed antiemetics.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toby Weingarten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Weingarten TN, McGlinch BP, Liedl L, Kendrick ML, Kellogg TA, Schroeder DR, Sprung J. Intranasal nicotine increases postoperative nausea and is ineffective in reducing pain following laparoscopic bariatric surgery in tobacco-Naive females: a randomized, double blind trial. Obes Surg. 2015 Mar;25(3):506-13. doi: 10.1007/s11695-014-1431-7. PMID 25190522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota from August 2010 to March 2014.
Pre-assignment Details: 95 subjects randomized; 48 to Placebo arm, and 47 to Nicotine arm. On the Placebo arm one subject had their surgery rescheduled and did not take part in the study, leaving 47 starting. On the Nicotine arm 3 subjects withdrew consent prior to surgery and 1 subject's surgery was cancelled, and 1 subject surgery rescheduled, leaving 42 starting.
Period: Overall Study
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray
Started | 42 | 47
Completed | 42 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray | Total
Number analyzed (Participants) | 42 | 47 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (9.1) | 44.9 (10.6) | 45.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 47 | 89

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Use During the Postanesthesia Care Unit (PACU) Stay, and the First 24 Hours Postoperatively
Description: Opioid use was calculated in intravenous morphine equivalents (iv MEQ) according to the Mayo Clinic Pharmacy opioid conversion calculator based on the recommendations from the American Pain Society. Specifically, the following conversion was used: 10 mg in MEQ=100mcg iv fentanyl=1.5 mg iv hydromorphone=20mg oral oxycodone=30mg oral hydrocodone.
Time Frame: During PACU stay (approximately 94 minutes after operation), 24 hours after operation
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray
Number analyzed (Participants) | 42 | 47
mg
  During the PACU stay | 5.3 [0 to 10.0] | 5.2 [0 to 12.7]
  First 24 hours postoperatively | 39.6 [20.0 to 52.5] | 32.7 [20.3 to 51.3]
Statistical Analysis 1: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; Comparison between arms for the postoperative opioid use during the postanesthesia care unit (PACU) stay, using a one tailed P value; Test type: Superiority or Other; p = 0.828, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; Comparison between the arms for the first 24 hours postoperatively, using a one tailed P value; Test type: Superiority or Other; p = 0.752, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants Who Needed to Use Antiemetic Medication in the PACU
Description: Rescue antiemetic therapy was 0.625 mg droperidol. Recalcitrant postoperative pain, nausea and vomiting (PONV) was treated per discretion of the supervising anesthesiologist.
Time Frame: 24 hours postoperatively.
Measure: Number; unit: participants
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray
Number analyzed (Participants) | 42 | 47
participants | 24 | 12
Statistical Analysis 1: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; Comparison between the arms for antiemetic medication use in the PACU; Test type: Superiority or Other; p = 0.002, Chi-squared

3. Secondary Outcome: Numeric Pain Score
Description: Upon arrival in the PACU and at least every 30 minutes thereafter while in the PACU, the subject was asked to report pain using a numerical pain score for current pain at rest from 0 (representing no pain) to 10 (representing the worst imaginable pain).
Time Frame: on admission, 30 minutes, 60 minutes, at discharge
Population: Not all participants completed the pain scale at every time point. The participants analyzed per arm (nicotine, normal) at each time point were: on admission (40, 45); 30 minutes (40, 47); 60 minutes (34, 40); at discharge (39, 44),
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray
Number analyzed (Participants) | 40 | 47
units on a scale
  On admission | 0 [0 to 6] | 3 [0 to 6]
  30 minutes | 5 [0.5 to 6] | 5 [0 to 7]
  60 minutes | 4 [2 to 6] | 4 [3 to 5]
  At discharge | 3 [2 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; The arms were compared for numeric pain score on admission; Test type: Superiority or Other; p = 0.354, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; The arms were compared for numeric pain score at 30 minutes; Test type: Superiority or Other; p = 0.492, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; The arms were compared for numeric pain score at 60 minutes; Test type: Superiority or Other; p = 0.809, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Nasal Nicotine Spray vs Nasal Normal Saline Spray; The arms were compared for numeric pain score at discharge; Test type: Superiority or Other; p = 0.381, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Nasal Nicotine Spray | Nasal Normal Saline Spray
Serious Adverse Events (participants affected / at risk) | 2/42 | 1/47
Other Adverse Events (participants affected / at risk) | 28/42 | 24/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Nicotine Spray (N=42) | Nasal Normal Saline Spray (N=47)
Anastomotic leak (Surgical and medical procedures) | 1 (1) | 0 (0) — An anastomotic leak is a breakdown along an anastomosis which causes fluids to leak. Anastomoses are used when a hollow organ needs to be severed and reconnected to allow fluids to flow through it.
Readmission for postoperative pain, nausea, and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Nicotine Spray (N=42) | Nasal Normal Saline Spray (N=47)
Postoperative pain, nausea, and vomiting (PONV) (Gastrointestinal disorders) | 27 (27) | 24 (24) — PONV was defined as any nausea score >0, use of rescue medication, or visible retching or vomiting.
Nasal burning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — At the end of 24 hours after the operation subjects were queried for the presence of nasal burning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes